CLINICAL TRIAL: NCT00640848
Title: Multi-center, Multiple-stage, Double-blind, Randomized, Placebo-controlled, Two-way Crossover, Single-dose Study to Investigate the Effects of ACT-078573 on Sleep Measured by Polysomnography in Patients With Primary Insomnia
Brief Title: Almorexant in Primary Insomnia
Acronym: Insomnia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Midnight Pharma, LLC (Industry)
Responsible Party: Jasper Dingemanse, Actelion
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-057-103
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Insomnia; Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — almorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: almorexant
- 2 (Experimental)
  Interventions: Drug: almorexant
- 3 (Experimental)
  Interventions: Drug: almorexant
- 4 (Experimental)
  Interventions: Drug: almorexant
- 5 (Experimental)
  Interventions: Drug: almorexant

INTERVENTIONS:
Drug: almorexant — 1 dose of 400 mg in two treatment sequences
  Other Names: ACT-078573
  Arms: 1
Drug: almorexant — 1 dose of 200 mg in two treatment sequences
  Other Names: ACT-078573
  Arms: 2
Drug: almorexant — 1 dose of 100 mg in two treatment sequences
  Other Names: ACT-078573
  Arms: 3
Drug: almorexant — 1 dose of 50 mg mg in two treatment sequences
  Other Names: ACT-078573
  Arms: 4
Drug: almorexant — 1 dose of 1000 mg in two treatment sequences
  Other Names: ACT-078573
  Arms: 5

SUMMARY:
The aim of the study is to determine the minimum effective dose of ACT-078573 on sleep efficiency and to assess the effects of different doses of ACT-078573 on other PSG parameters.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 - 65 years of age (inclusive).
* Women of childbearing potential must have a negative urine pregnancy test at the screening visit, the screening adaptation night, and pre-treatment and use a reliable method of contraception during the entire study duration and for at least 3 months after study drug intake.

Reliable methods of contraception are:

* Barrier type devices (e.g., female condom, diaphragm, contraceptive sponge) only in combination with a spermicide.
* Intra-uterine devices.
* Oral, injectable, implantable or transdermal contraceptives only in combination with a barrier method.

  * Abstention, rhythm method, and contraception by the partner alone are not acceptable methods of contraception.

Women not of childbearing potential are defined as prepubescent, postmenopausal (i.e., amenorrhea for at least 1 year), or surgically or naturally sterile.

* Body mass index (BMI) between 18 and 30 kg/m2 (limits included) at screening visit.
* 12-lead ECG without clinically relevant abnormalities at screening visit.
* Hematology and biochemistry test results not deviating from the normal range to a clinically relevant extent at screening visit and following the screening/adaptation night.
* Primary insomnia by DSM-IV-TR criteria based on medical history and the assessments performed at screening visit.
* History of the following for at least 3 months prior to the screening visit:

  * Usual reported subjective total sleep time (TST) 3 - 6 hours.
  * Usual sleep disturbance with a subjective sleep onset latency of > 30 min.
  * Daytime complaints associated with poor sleep (e.g., fatigue, irritability, difficulty concentrating).
* Polysomnography (PSG) at screening/adaptation night confirming TST < 6 h and LPS ≥ 20 min.
* Willingness to refrain from CNS-active drugs for 5 half-lives of the respective drug (but at least 1 week) prior to the screening/adaptation night and up to the end of treatment period 2. The usage of short-acting hypnotics (defined as hypnotics with a half-life of up to and including 10 hours) is allowed up to 48 hours prior to each PSG night, i.e., prior to the screening/adaptation night and prior to the treatment PSG nights.
* Urine drug test negative for barbiturates, cannabinoids, amphetamines, and cocaine at screening visit 1, screening/adaptation PSG night and pre-treatment. Urine drug test negative for benzodiazepines and opiates at screening/adaptation PSG night and pre-treatment.
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Symptom assessment questionnaire (SBB) for diagnosis of apnea resulting in a score > 2 at screening visit.
* Zung self-rating depression scale (SDS) and/or Zung self-rating anxiety scale (SAS) resulting in a raw score ≥ 50 at screening visit.
* Restless legs syndrome and/or meeting all four essential diagnostic criteria for RLS (see Appendix 10).
* Insomnia due to sleep apnea or periodic limb movement disorder as assessed by PSG at screening/adaptation night:

  * apnea/hypopnea index (AHI) > 10/h
  * periodic limb movement arousal index > 10/h
* Major depressive disorder, severe psychosis, or significant anxiety disorder.
* Pregnancy or breast-feeding.
* Systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg at screening visit.
* Within the 2-month period prior to the screening visit, clinical evidence of alcoholism or drug abuse.
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as psychiatric disease or a disease which may affect the pharmacokinetics of the study drug.
* Treatment with strong inhibitors of CYP3A4 (e.g., azole derivatives, ritonavir, clarithromycin) within 1 week prior to the screening/adaptation PSG night and up to the end of treatment period 2.
* Excessive caffeine consumption (regular caffeine consumption of > 7 units per day).
* Night shift workers.
* Known hypersensitivity to any excipients of the drug formulation.
* Planned treatment or treatment with another investigational drug within 1 month prior to randomization and up to the end of treatment period 2.
* Known concomitant life-threatening disease with a life expectancy < 24 months.
* Unstable medical abnormality, significant medical disorder or acute illness.
* Recruitment of the same patient twice to the same dose level. Patients may be recruited to a lower dose level, provided that there are at least 28 days between last study drug administration and screening/adaptation PSG night.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency (%) assessed by PSG (polysomnography) | Between 10pm-12am (=lights out) until 480 minutes thereafter (=lights on)

SECONDARY OUTCOMES:
LPS (Latency to Persistent Sleep) [min] assessed by PSG (polysomnography) | Time from start of recording to the beginning of the first continuous 20 epochs of non-wake

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Dingemanse, PhD, Study Director — Actelion; Eleornora Chiossi, MSc, Study Director — Actelion; Petra Hoever, MSc, Study Director — Actelion; Fabrice Kramer, MD, Study Director — Actelion; Georg Dorffner, Prof. Dr., Principal Investigator — The Siesta Group
Locations (27):
- Austria (4):
  - Medical University of Innsbruck, Dept. of Neurology Sleep Disorder Unit, Innsbruck
  - Medical University of Vienna, Clinic of Neurology, Vienna
  - Medical University of Vienna, University Clinic of Psychiatrie, Vienna
  - The Siesta Group, Vienna
- Denmark (2):
  - Scan Sleep, Copenhagen
  - Glostrup University Hospital Department of Sleep Medicine, Glostrup Municipality
- Finland (2):
  - Skogby Sleep Clinic, Espoo
  - Sleep Research Unit, Dentalia, University of Turku, Turku
- Germany (8):
  - Charite Campus Benjamin Franklin, Klinik und Hochschulambulanz fur Psychiatrie and Psychotherapie, Berlin
  - Department of Internal Medicine, Center for Sleep Medicine, Berlin
  - St Hedwig-Krankenhaus, Akademisches Lehrkrankenhaus der Charite, Berlin
  - Department of Psychiatry and Psychotherapy of the University Hospital of Freiburg, Freiburg im Breisgau
  - St. Valentinushaus Klinik fur Psychiatrie und Psychotherapie, Kiedrich
  - Universitatsklinikum Giessen und Marburg, Standort Marburg, Nervenklinik, Marburg
  - Klinik und Poliklinik fur Psychiatrie, Psychosomatik und Psychotherapie der Universitat am Bezirsklinikum, Regensburg
  - SOMNIBENE Institut fur Medzinische Forschung und Schlafmedizin, Schwerin
- Israel (2):
  - Technion Sleep Medicine Center, Rambam Medical Center, Haifa
  - Assuta Medical Centers, Petah Tikva
- Medisch Centrum Haaglanden-Westeinde Ziekenhuis, Slaapcentrum (Holland Sleep Research), The Hague, Netherlands
- Spain (2):
  - Hospital de la Ribera, Alzira
  - Hospital de la Santa Crue/Sant Pau, Institut de Recerca, Barcelona
- Sweden (2):
  - Skaraborg Hospital, Sleep Medicine Unit, Department of Neurorehabilitation, Skövde
  - Uppsala Akademiska Hospital, Sleep Disorder Unit, Uppsala
- Switzerland (2):
  - Psychiatric University Clinics (UPK) Basel, Dept. for Depression Research, Sleep Medicine and Neurophysiology, Basel
  - University Hospital Zurich (USZ), Neurology Polyclinic, Center for Sleep Medicine, Zurich
- United Kingdom (2):
  - The Edinburgh Sleep Centre, Edinburgh
  - Medical Director, The London Sleep Centre, London

REFERENCES:
- [Derived] Hoever P, Dorffner G, Benes H, Penzel T, Danker-Hopfe H, Barbanoj MJ, Pillar G, Saletu B, Polo O, Kunz D, Zeitlhofer J, Berg S, Partinen M, Bassetti CL, Hogl B, Ebrahim IO, Holsboer-Trachsler E, Bengtsson H, Peker Y, Hemmeter UM, Chiossi E, Hajak G, Dingemanse J. Orexin receptor antagonism, a new sleep-enabling paradigm: a proof-of-concept clinical trial. Clin Pharmacol Ther. 2012 Jun;91(6):975-85. doi: 10.1038/clpt.2011.370. PMID 22549286